CLINICAL TRIAL: NCT01374191
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Crossover Clinical Trial of Botulinum Toxin Type A for Neuroma Pain
Brief Title: Botulinum Toxin Type A for Neuroma Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-SIUSOM-11-002
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Neuroma
Keywords: botox; neuroma pain; pain; chronic pain; botulinum toxin; botulinum toxin A; botox and pain; botox and neuroma; botox treatment; onabotulinum; onabotulinum toxin; onabotulinum toxin type A
MeSH Terms: conditions — Neuroma; Pain; Chronic Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- onabotulinum toxin type-A (Active Comparator): 1 injection of Btx-A, or up to 4 injections of Btx-A during the 1-year study period if pain recurs
  Interventions: Drug: onabotulinum toxin type-A
- placebo (Placebo Comparator): saline
  Interventions: Other: placebo
- 2nd phase - onabotulinum toxin type-A (Active Comparator): 2 - 3 injections of Btx-A, specific to patient pain recurrence
  Interventions: Drug: 2nd phase - onabotulinum toxin type-A

INTERVENTIONS:
Drug: onabotulinum toxin type-A — 1 injection of Btx-A
  Other Names: Botulinum Toxin Type A; Botox
  Arms: onabotulinum toxin type-A
Other: placebo — 1 injection of saline solution
  Arms: placebo
Drug: 2nd phase - onabotulinum toxin type-A — 2 - 3 injections of Btx-A, specific to patient pain recurrence
  Other Names: Botulinum Toxin Type A; Botox
  Arms: 2nd phase - onabotulinum toxin type-A

SUMMARY:
The purpose of this study is to determine if botulinum toxin type A (Btx-A) is an effective treatment for painful neuromas. The ideal therapy for painful neuromas would be effective, non-addictive, safe, localized, and cost-effective treatment. At the same time, the therapy would also address the complex peripheral and central mechanisms. Btx-A is a potential treatment that addresses each of these requirements while preserving the existing sensation and function.

Study Hypothesis: Btx-A injection relieves neuroma pain better than a placebo

DETAILED DESCRIPTION:
PROJECT SUMMARY OVERVIEW: The purpose of this study is to determine if botulinum toxin type A (Btx-A) is an effective treatment for painful neuromas. The ideal therapy for painful neuromas would be effective, non-addictive, safe, localized, and cost-effective, but would also address the complex peripheral and central mechanisms. Btx-A is a potential treatment that addresses each of these requirements while preserving the existing sensation and function. The investigators believe that Btx-A will be effective in eliminating both the exaggerated local pain response and centralization while maintaining an exceptional safety profile and potential for long-term effects without addictive properties.

STUDY AIMS: The aims of this proposal are to 1) examine the short-term efficacy of Btx-A injection compared to placebo in treating pain due to nerve damage, and 2) describe the long-term efficacy of Btx-A injection in treating pain due to nerve damage by measuring patient satisfaction and quality of life changes over time.

APPROACH: Forty patients will be enrolled; twenty to receive active treatment (Btx-A) and twenty to receive placebo (saline). Comparisons between treatment and placebo will occur during the first 28 days to determine Btx-A's short-term efficacy. Telephone follow-up visits will occur on Day 2 and Week 1. On Day 28, a telephone follow-up visit will occur, except in patients who are experiencing complications. Patients with complications or recurrent pain will return for a clinic visit. Post-assessment on Day 28 marks the beginning of the longitudinal observational study of patient outcomes. Placebo will no longer be used and patients still suffering from pain will be eligible for additional Btx-A injections. Patients may receive up to 4 injections of Btx-A during the 1-year study period if pain recurs. During the study period participants will be followed to collect data on pain-free intervals, subsequent treatment choices, patient satisfaction, and changes in quality of life and function. Group comparisons will be made to analyze results. Further stratifications for data analysis will be made as enrollment numbers allow to control for additional demographic and disease variables. Quality-adjusted life-years will be calculated to help determine the societal and individual cost of this treatment.

HYPOTHESIS: The investigators hypothesize that 1) Btx-A injection relieves neuroma pain better than a placebo within 28 days of injection, and 2) Btx-A injection relieves neuroma pain for longer than 28 days, improving patient quality of life. Through this study the investigators intend to further elucidate the efficacy of injected Btx-A on relieving chronic pain from nerve damage while characterizing the patients for whom this treatment is most effective.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* aged 18-75 years
* diagnosed with neuroma pain
* able to return/be available for follow-up evaluations
* willingness and ability to give informed consent

Exclusion Criteria:

* positive for HIV/AIDS or otherwise immunocompromised
* history of neuromuscular disease
* reported allergy to BOTOX®
* history or symptoms of any significant medical problem in the last year (i.e., bradycardia, impaired cardiovascular function, liver disease)
* symptoms of infection or illness with initial enrollment
* pregnant or lactating women
* unable or unwilling to maintain abstinence or use contraception for 28 days following all injections
* cognitively impaired patients unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
number of pain-free days | change from baseline to 28 days
  subjective evaluation of pain relief, using Subjective pain scales [visual analogue scale (VAS) and faces pain assessment]

SECONDARY OUTCOMES:
quality of life | change from baseline to 28 days
  SF-12v2® Health Survey - Pain Enhanced
upper extremity function | change from baseline to 28 days
  Quick-DASH (Disabilities of the Arm, Shoulder, and Hand) Outcome Measure
lower extremity function | change from baseline to 28 days
  Lower Extremity Functional Scale (LEFS)
patient satisfaction | change from baseline to 28 days
  SF-12v2® Health Survey - Pain Enhanced
quality-adjusted life-years | change from baseline to 28 days
  EuroQol (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Neumeister, MD, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- [Background] Neumeister MW. Botulinum toxin type A in the treatment of Raynaud's phenomenon. J Hand Surg Am. 2010 Dec;35(12):2085-92. doi: 10.1016/j.jhsa.2010.09.019. PMID 21134617
- [Background] Neumeister MW, Chambers CB, Herron MS, Webb K, Wietfeldt J, Gillespie JN, Bueno RA Jr, Cooney CM. Botox therapy for ischemic digits. Plast Reconstr Surg. 2009 Jul;124(1):191-201. doi: 10.1097/PRS.0b013e3181a80576. PMID 19568080
- See also: U.S. Food & Drug Administration webpage on drugs with consumer information links — http://www.fda.gov/Drugs/default.htm
- See also: U.S. Food and Drug Administration search page for FDA approved drug products — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.DrugDetails